CLINICAL TRIAL: NCT04699279
Title: Protective Effect of Statin Against Negative Cardiovascular Remodeling and Organ Dysfunction After Acute Aortic Syndrome Surgery (PANDA III)
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); West China Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The Affiliated Hospital of Qingdao University Medical College (Unknown)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular surgery Dept., Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PANDA III
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acute Aortic Syndrome; Aortopathy
MeSH Terms: conditions — Acute Aortic Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin (Experimental)
  Interventions: Drug: Rosuvastatin 10mg
- Blank (No Intervention)

INTERVENTIONS:
Drug: Rosuvastatin 10mg — Rosuvastatin 10mg is taken by oral or nasal feeding every day at ang time.
  Arms: Statin

SUMMARY:
Acute Aortic Syndrome (AAS)/Aortic Aneurysm is a common feature of aortic wall events, including aortic dissection, intramural hematoma, aortic ulceration and aortic trauma, and occurs in up to 35 cases per 100,000 cases per year between the ages of 65 and 75 years. Increased levels of the inflammatory biomarker high-sensitivity C-reactive protein predict cardiovascular events. Since statins lower levels of high-sensitivity C-reactive protein as well as cholesterol, the authors hypothesized that people with acute aortic syndrome but without hyperlipidemia might benefit from statin treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with aortic dissection/ulceration/intermural hematoma/aortic aneurysm who underwent aortic arch replacement or endoluminal isolation or hybrid therapy;
* (2) Paitents without clinically significant hyperlipidemia but with cardiovascular disease risk factors (such as male ≥45 years old, female ≥55 years old, hypertension, diabetes, chronic kidney disease, obesity, low HDL cholesterol, smoking, alcohol consumption, family history of early onset ischemic cardiovascular disease) and no previous use of statins;
* (3) Patients are between 18 and 85 years old, male or female;
* (4) Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* (1) Patients with allergy to statins;
* (2) patients with active liver disease;
* (3) patients with myopathy;
* (4) Lactating women and pregnant women;
* (5) Patients with mental diseases, drug and alcohol dependence;
* (6) Refuse to participate in the study or sign the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Aortic adverse events | 3 months after surgery
  a composite outcomes event of aortic rupture, aortic dissection, severe dilation of the aorta, and cardiac death.

SECONDARY OUTCOMES:
Mortality | 3 months after surgery
  Death from any cause

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Beijing Anzhen Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided